CLINICAL TRIAL: NCT06443385
Title: E-mails to Nudge Safer and Better-Informed Prescribing of Risky Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Southern California (Other); Bowdoin College (Other); Abdul Latif Jameel Poverty Action Lab (Other); Minnesota Management and Budget (Unknown); Minnesota Board of Pharmacy (Other)
Responsible Party: Principal Investigator, Adam Sacarny, PhD, Associate Professor of Health Policy and Management, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAV1928; AEARCTR-0013549 (Registry Identifier: AEA RCT Registry (socialscienceregistry.org))
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Opioid Prescribing; Prescription Drug Misuse
Keywords: opioids; prescribing; overprescribing; prescription drug monitoring programs; controlled substances
MeSH Terms: conditions — Prescription Drug Misuse

STUDY DESIGN:
Intervention Model Description: Clinicians will be assigned at random to one of three arms: PDMP legal mandate e-mails, PDMP clinical benefit emails, or a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Legal Mandate Messaging (Experimental)
  Interventions: Behavioral: PDMP Legal Mandate E-mail
- Clinical Benefit Messaging (Experimental)
  Interventions: Behavioral: PDMP Clinical Benefit E-mail
- Control (No Intervention)

INTERVENTIONS:
Behavioral: PDMP Legal Mandate E-mail — E-mails highlighting the state's legal requirements to use the PDMP. There will be one initial email and one follow-up email one month later.
  Arms: Legal Mandate Messaging
Behavioral: PDMP Clinical Benefit E-mail — E-mails highlighting the clinical benefits of having access to the PDMP and checking the PDMP before prescribing opioids. There will be one initial email and one follow-up email one month later.
  Arms: Clinical Benefit Messaging

SUMMARY:
This study will test e-mails to encourage engagement with the Minnesota prescription monitoring program (PMP/PDMP) and will evaluate the effect of these e-mails on PMP/PDMP use and controlled substance prescribing.

DETAILED DESCRIPTION:
Drug overdose deaths have skyrocketed in recent years, and many overdoses continue to involve prescribed medications like opioids and stimulants. At the same time, state prescription drug monitoring programs (PDMPs), which help clinicians prescribe these medications safely, remain underused. In Minnesota, 32% of opioid prescriptions are written by clinicians who do not use the PDMP. In many states, including Minnesota, policymakers have limited tools to raise PDMP use even though it is often required under state law. To address this policy dilemma, this study will test e-mails designed to facilitate PDMP use and evaluate their effects on PDMP use and controlled substance prescribing. This study will include a projected 7,126 physician and physician assistant prescribers of opioids and other controlled substances who lack active PDMP accounts, never query the PDMP, or query the PDMP infrequently relative to their prescribing volume. To generate evidence on clinician motivation for responding to encouragement, the study will randomly vary messaging to focus on legal requirements to use the PDMP vs. clinical benefits of the PDMP.

ELIGIBILITY:
Inclusion Criteria:

* Minnesota physician or physician assistant
* Controlled substance prescriber not following state requirements to maintain an active PDMP account, or opioid prescriber not searching the PDMP or infrequently searching the PDMP

Exclusion Criteria:

* No e-mail address available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7872 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Rate of PDMP Engagement | 2 months
  An indicator for increased PDMP engagement during the 2-month period after the first e-mails were sent. It will indicate whether the level of engagement rose from the baseline level that resulted in the clinician's enrollment into the study. For clinicians who lacked an account, the outcome will indicate whether they created one; for clinicians with an inactive account, the outcome will indicate whether they reactivated it. For those who never searched, it will indicate any search, and for those who rarely searched, it will indicate whether their search rate rose.
Volume of Potentially Guideline-discordant Opioid Prescribing | 2 months
  A composite of several measures of potentially guideline-discordant opioid prescribing. These will include:
  1. Opioid co-prescriptions with other opioids
  2. Opioid co-prescriptions with benzodiazepines
  3. Opioid co-prescriptions with gabapentinoids
  4. High daily opioid doses
  5. Long-duration opioid prescriptions to opioid-naïve individuals

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sacarny, PhD, Principal Investigator — Columbia University; Mireille Jacobson, PhD, Principal Investigator — University of Southern California; Tatyana Avilova, PhD, Principal Investigator — Bowdoin College
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sacarny A, Avilova T, Williamson I, Merrick W, Jacobson M. Prescription Drug Monitoring Program Reminder Emails, Program Use, and Prescribing: A Randomized Clinical Trial. JAMA Health Forum. 2025 Dec 5;6(12):e255623. doi: 10.1001/jamahealthforum.2025.5623. PMID 41632198